CLINICAL TRIAL: NCT01921751
Title: A Phase II Randomized Trial Evaluating the Addition of High or Standard Intensity Radiation to Gemcitabine and Nab-paclitaxel for Locally Advanced Pancreatic Cancer
Brief Title: High or Standard Intensity Radiation Therapy After Gemcitabine Hydrochloride and Nab-paclitaxel in Treating Patients With Pancreatic Cancer That Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial would not be completed in a reasonable timeframe per CTEP guidelines
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 1201; NCI-2013-01280 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RTOG 1201 (Other: NRG Oncology); RTOG-1201 (Other: CTEP); U10CA180868 (NIH); U10CA021661 (NIH)
Record Dates: First submitted 2013-08-09; First posted 2013-08-13 (Estimated); Results first posted 2018-03-22 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-06

CONDITIONS: Pancreatic Adenocarcinoma; Stage III Pancreatic Cancer
Keywords: SMAD4; IMRT; gemcitabine; high-dose radiotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Capecitabine; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Chemotherapy + high intensity radiation (Experimental): Induction chemotherapy with four cycles of gemcitabine and nab-paclitaxel [randomized to this arm after 3rd cycle and no progression]; followed by concurrent high intensity radiation therapy and capecitabine; followed by consolidation chemotherapy with gemcitabine and nab-paclitaxel until progression or unacceptable toxicity
  Interventions: Drug: Capecitabine; Drug: Gemcitabine; Radiation: high intensity radiation therapy; Drug: nab-Paclitaxel
- Chemotherapy + low intensity radiation (Experimental): Induction chemotherapy with four cycles of gemcitabine and nab-paclitaxel [randomized to this arm after 3rd cycle and no progression]; followed by concurrent low intensity radiation therapy and capecitabine; followed by consolidation chemotherapy with gemcitabine and nab-paclitaxel until progression or unacceptable toxicity
  Interventions: Radiation: low intensity radiation therapy; Drug: Capecitabine; Drug: Gemcitabine; Drug: nab-Paclitaxel
- Chemotherapy (Active Comparator): Gemcitabine and nab-paclitaxel until progression or unacceptable toxicity [randomized to this arm after 3rd cycle and no progression]
  Interventions: Drug: Gemcitabine; Drug: nab-Paclitaxel

INTERVENTIONS:
Radiation: low intensity radiation therapy — 50.4 Gy in 28 1.8 Gy fractions (IMRT or 3D-CRT), 5 days/week, starting 3-5 weeks after the last dose of induction chemotherapy
  Other Names: 3-dimensional conformal radiation therapy; 3-dimensional radiation therapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; IMRT; intensity modulated radiation therapy; intensity-modulated radiation therapy; Intensity-Modulated Radiotherapy; Intensity Modulated RT
  Arms: Chemotherapy + low intensity radiation
Drug: Capecitabine — 825 mg/m2 PO twice daily, 5 days/week, beginning on the first day of radiation therapy and ending on the last day of radiation therapy.
  Other Names: Ro 09-1978/000; Xeloda
  Arms: Chemotherapy + high intensity radiation; Chemotherapy + low intensity radiation
Drug: Gemcitabine — 1000 mg/m2 weekly as a 30 minute infusion after nab-Paclitaxel, three weeks on and 1 week off [1 cycle = 4 weeks]
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; GEMCITABINE HYDROCHLORIDE; Gemzar; LY-188011
Radiation: high intensity radiation therapy — 63 Gy intensity-modulated radiation therapy (IMRT) in 28 2.25 Gy fractions, 5 days/week, starts 3-5 weeks after the last dose of induction chemotherapy
  Other Names: IMRT; Intensity Modulated RT; intensity-modulated radiation therapy; Intensity-Modulated Radiotherapy
  Arms: Chemotherapy + high intensity radiation
Drug: nab-Paclitaxel — 125 mg/m2 weekly as a 30-40 minute infusion, three weeks on and 1 week [1 cycle = 4 weeks]
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel

SUMMARY:
This randomized phase II trial studies how well high or standard intensity radiochemotherapy after gemcitabine hydrochloride and paclitaxel albumin-stabilized nanoparticle formulation (nab-paclitaxel) work compared with gemcitabine hydrochloride and nab-paclitaxel alone in treating patients with pancreatic cancer that cannot be removed by surgery. Drugs used in chemotherapy, such as gemcitabine hydrochloride and nab-paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs, such as capecitabine, may make tumor cells more sensitive to radiation therapy. Giving radiation therapy in different ways and adding chemotherapy may kill more tumor cells. It is not yet known whether high intensity radiochemotherapy after gemcitabine hydrochloride and nab-paclitaxel is more effective than standard intensity radiochemotherapy after gemcitabine hydrochloride and nab-paclitaxel or gemcitabine hydrochloride and nab-paclitaxel alone in treating pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* I. To determine if intensified radiochemotherapy following gemcitabine and nab-paclitaxel in patients with unresectable pancreatic cancer will show a signal for improved 2-year overall survival (OS) from 10% to 22.5% as compared to chemotherapy with gemcitabine and nab-paclitaxel alone.
* II. To determine if standard radiochemotherapy, following gemcitabine and nab-paclitaxel, in patients with unresectable pancreatic cancer will show a signal for improved 2-year OS from 10% to 22.5% as compared to chemotherapy with gemcitabine and nab-paclitaxel alone.

SECONDARY OBJECTIVES:

* I. To evaluate patterns of failure (local and systemic progression) by SMAD family member 4 (SMAD4) status and intensity of radiation therapy.
* II. To evaluate the impact of radiochemotherapy on OS for the subset of SMAD4 intact patients.
* III. To evaluate adverse events associated with the treatments.
* IV. To evaluate correlation between SMAD4 status determined by immunohistochemistry (IHC) and genetic SMAD4 status.

Patients are randomized to 1 of 3 treatment arms.

After completion of study treatment, patients are followed up at 1 month and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven diagnosis of adenocarcinoma of the pancreas prior to registration
2. Tumor diameter ≤ 7 cm
3. Unresectable by radiographic criteria (pancreas protocol CT or MRI) or exploration within 30 days prior to registration.
4. A cell block or core biopsy must be submitted for central review and analysis of SMAD4 status as soon as possible following step 1 registration.
5. No distant metastases, based upon the following minimum diagnostic workup:

   * History/physical examination within 30 days prior to registration
   * Whole body fluorodeoxyglucose-positron emission tomography/computerized tomography (FDG-PET/CT) within 30 days prior to registration NOTE: If whole-body FDG-PET/CT is not performed, CT of the chest and CT (or MRI) of abdomen and pelvis must be obtained (imaging of abdomen and pelvis need not be repeated if already included in pancreas protocol study)
6. Zubrod Performance Status 0-1 within 30 days prior to registration
7. Age ≥ 18;
8. Complete blood count (CBC)/differential obtained within 14 days prior to step 1 registration, with adequate bone marrow function defined as follows:

   * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
   * Platelets ≥ 100,000 cells/mm3
   * Hemoglobin ≥ 8.0 g/dl (NOTE: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable)
9. Additional laboratory studies within 14 days prior to registration:

   * carbohydrate antigen 19-9 (CA19-9); NOTE: in the event that a stent has been placed and biliary obstruction has been relieved, the CA19-9 should be drawn post stent placement
   * Creatinine < 2 mg/dl; Glomerular filtration rate (GFR) > 50 mL/min (Cockroft and Gault formula)
   * Bilirubin < 1.5 x ULN
   * Alanine aminotransferase (ALT) and aminotransferase (AST) ≤ 2.5 x ULN
   * Activated partial thromboplastin time (aPTT), prothrombin time (PT) ≤1.2 x upper limit of normal (ULN)
10. Patient must provide study specific informed consent prior to study entry
11. Women of childbearing potential and male participants must practice adequate contraception during protocol treatment and for at least 6 months following treatment
12. For females of child-bearing potential, negative serum pregnancy test within 30 days prior to registration

Exclusion Criteria:

1. More than one primary lesion
2. Prior invasive malignancy (unless disease free for a minimum of 1095 days [3 years]); Non-melanomatous skin cancer and previous early prostate cancer that had a non-rising prostate-specific antigen (PSA) are eligible
3. Prior systemic anti-cancer therapy for pancreatic cancer; note that prior chemotherapy for a different cancer is allowable
4. Prior radiation therapy to the abdomen that would result in overlap of radiation therapy fields
5. Severe, active co-morbidity, defined as follows:

   * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
   * Transmural myocardial infarction within the last 6 months
   * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
   * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration
   * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol
   * Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients
6. Pregnancy or women of childbearing potential, women who cannot discontinue breastfeeding and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
7. Prior allergic reaction to the study drug(s) involved in this protocol
8. Pre-existing Grade 2 or greater neuropathy
9. Distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Ben-Josef, Principal Investigator — NRG Oncology
Locations (46):
- United States (46):
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Saint Joseph Hospital, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - OSF Saint Francis Medical Center Radiation Oncology Service at the Central Illinois Comprehensive CC, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - University of Rochester, Rochester, New York
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Door County Cancer Center, Sturgeon Bay, Wisconsin

REFERENCES:
- [Derived] Jani A, Horowitz DP. Radiation Therapy Deviations in Trial of Locally Advanced Pancreatic Cancer [corrected]. JAMA. 2016 Oct 4;316(13):1409. doi: 10.1001/jama.2016.9778. No abstract available. PMID 27701653

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were registered and received 3 cycles of Gemcitabine/nab-Paclitaxel and then had central SMAD4 testing done. Patients then had a CT/MRI of their abdomen/pelvis for restaging. Only non-progressing patients were then randomized after being stratified by carbohydrate antigen 19-9 (CA19-9) and SMAD4.
Period: Overall Study
Arm/Group | Chemotherapy + High Intensity Radiation | Chemotherapy + Low Intensity Radiation | Chemotherapy
Started | 4 | 4 | 5
Completed | 4 (All randomized patients are reported here.) | 4 (All randomized patients are reported here.) | 5 (All randomized patients are reported here.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy + High Intensity Radiation | Chemotherapy + Low Intensity Radiation | Chemotherapy | Total
Number analyzed (Participants) | 4 | 4 | 5 | 13
Age, Continuous [Median (Full Range); unit: years] | 63.5 [62 to 69] | 69 [59 to 71] | 66 [60 to 68] | 66 [59 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 9
  Male | 0 | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Survival time is defined as time from randomization to date of death from any cause and was to be estimated by the Kaplan-Meier method. Given the limited follow-up due to early closure and termination of data collection, only the number of patients last reported to be alive at time of study termination is reported.
Time Frame: From randomization until last follow-up. Analysis was to occur after a total of 140 deaths were reported within the pairing of each radiation arm with the chemotherapy alone arm. Maximum follow-up at time of study termination was 8.3 months.
Population: All randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy + High Intensity Radiation | Chemotherapy + Low Intensity Radiation | Chemotherapy
Number analyzed (Participants) | 4 | 4 | 5
Participants | 4 | 4 | 5

2. Secondary Outcome: Overall Survival Within SMAD4 Subsets
Description: Survival time is defined as time from randomization to date of death from any cause and was to be estimated by the Kaplan-Meier method. Given the limited follow-up due to early closure and termination of data collection, only the number of patients last reported to be alive at time of study termination is reported. Patients are categorized by SMAD4 status of "intact" (positive nuclear labeling is observed of the neoplastic cells ), "loss" (no labeling observed of the neoplastic cells) , or "undetermined" (insufficient material for immunostaining or results are equivocal). This study terminated early with only 20 registered (346 planned) and 13 randomized (288 planned). There are no proven results as to which category has better incomes, but this study hypothesizes that "intact" is highly correlated with local failures and "loss" is highly correlated with widespread metastasis, in which case "intact" would correspond with positive results relative to "loss".
Time Frame: as for outcome 1
Population: All randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy + High Intensity Radiation | Chemotherapy + Low Intensity Radiation | Chemotherapy
Number analyzed (Participants) | 4 | 4 | 5
Participants
  Intact | 1 | 1 | 3
  Loss | 3 | 2 | 1
  Undetermined | 0 | 1 | 1

3. Secondary Outcome: Patterns of Failure (Local and Metastatic Failure)
Description: Local progression is defined as least a 20% increase in the sum of diameters of the primary, taking as reference the baseline sum. Given the inherent inaccuracy in determining size of a primary pancreatic carcinoma, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm and progression must be demonstrated on at least two sequential scans. Metastatic failure is defined as metastatic disease. Local and distant failure were to be estimated by the cumulative incidence method. Given the limited follow-up due to early closure and termination of data collection, only the number of patients with failure is reported.
Time Frame: From randomization until last follow-up. Maximum follow-up at time of study termination was 8.3 months.
Population: Randomized eligible patients with follow-up data.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy + High Intensity Radiation | Chemotherapy + Low Intensity Radiation | Chemotherapy
Number analyzed (Participants) | 1 | 2 | 0
Participants
  Local Failure | 0 | 0 |
  Metastatic Failure | 0 | 1 |

4. Secondary Outcome: Correlation Between SMAD4 Status Determined by Immunohistochemistry (IHC) and Genetic SMAD4 Status
Time Frame: Baseline
Population: Because the study was terminated early, genetic SMAD4 status was not determined and therefore this analysis will not occur.
Arm/Group | Chemotherapy + High Intensity Radiation | Chemotherapy + Low Intensity Radiation | Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: Registered patients with adverse event data are included. Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Groups:
- Chemotherapy - Not Randomized: Induction chemotherapy with three cycles of gemcitabine and nab-paclitaxel [not randomized]
Arm/Group | Chemotherapy + High Intensity Radiation | Chemotherapy + Low Intensity Radiation | Chemotherapy | Chemotherapy - Not Randomized
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/4 | 1/5 | 1/7
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 5/5 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + High Intensity Radiation (N=4) | Chemotherapy + Low Intensity Radiation (N=4) | Chemotherapy (N=5) | Chemotherapy - Not Randomized (N=7)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Edema limbs (General disorders) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell decreased (Investigations) | 1 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + High Intensity Radiation (N=4) | Chemotherapy + Low Intensity Radiation (N=4) | Chemotherapy (N=5) | Chemotherapy - Not Randomized (N=7)
Anemia (Blood and lymphatic system disorders) | 4 | 2 | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0
Blurred vision (Eye disorders) | 2 | 0 | 0 | 1
Eye disorders - Other, specify (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 2 | 1
Bloating (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 3 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 1
Edema limbs (General disorders) | 1 | 1 | 0 | 0
Fatigue (General disorders) | 4 | 2 | 5 | 2
Fever (General disorders) | 1 | 0 | 0 | 1
Localized edema (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 2 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 1 | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 2 | 2
Alkaline phosphatase increased (Investigations) | 0 | 2 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 2
Lymphocyte count decreased (Investigations) | 1 | 2 | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 2 | 3 | 1
Platelet count decreased (Investigations) | 3 | 1 | 3 | 2
Weight gain (Investigations) | 0 | 1 | 0 | 0
Weight loss (Investigations) | 1 | 1 | 2 | 1
White blood cell decreased (Investigations) | 4 | 3 | 4 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 3 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 1
Dysesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2 | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 3 | 2 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Hot flashes (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 3 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0
Lymphedema (Vascular disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
This study terminated early with only 20 registered (346 planned) and 13 randomized (288 planned). Follow-up forms were collected on only 3 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.